CLINICAL TRIAL: NCT03692481
Title: Evolution of Lung 18FDG Uptake in Patients With Idiopathic Pulmonary Fibrosis and Receiving Pirfenidone
Acronym: PET-Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P180301J
Record Dates: First submitted 2018-09-14; First posted 2018-10-02 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis (IPF); 18FDG uptake; prognosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18FDG-PET scan (Experimental): 18FDG PET scan will be performed in each patient before initiation of pirfenidone and after 12 weeks of treatment
  Interventions: Radiation: 18FDG-PET scan

INTERVENTIONS:
Radiation: 18FDG-PET scan — 18FDG PET scan will be performed in each patient before initiation of pirfenidone and after 12 weeks of treatment

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a rare and fatal lung disease characterized by unpredictable changes with variable kinetics of progression. Changes in pulmonary function (FVC, DLCO) assessed at the time of diagnosis, or decline in pulmonary function within 12 months after diagnosis, are the best predictors of survival, but poorly predicted disease activity and evolution. 18FDG positron emission tomography (18FDG PETscan) provides the ability to quantify cell metabolism in vivo and non-invasively using a labeled non-metabolizable substrate. Several parameters can be measured in an automated and reproducible way, such as the mean fixation intensity (SUV mean), the maximum fixation intensity (SUV max), the hyperfixing volume measurement (MLV) or the glycolytic activity measurement tissue or TLG (total lesions glycolysis). Several studies have demonstrated an increase of glycolytic activity in lung fibroblast from IPF patient. In a recent study, the investigators demonstrated a strong correlation between the lung uptake parameters and the lung function tests results (LFTs) and prognostic score GAP. In addition, MLV and TLG were factors prognostic and independently associated with progression-free survival at 12 months. In a preliminary study, the investigators studied the change of these parameters in twelve patients treated with pirfenidone for IPF who performed an 18FDG PETscan before the initiation of treatment and about twelve weeks later. A mean decrease of 30% in TLG value between the two evaluations was observed. These preliminary data suggest that pirfenidone influences lung metabolism in patients with IPF. The investigators aim to conduct a prospective study to confirm and refine the preliminary data.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a rare and fatal lung disease characterized by an unpredictable evolution with variable kinetics of progression and burdened by the occurrence of exacerbation. The evaluation of the prognosis in a given patient remains difficult. Impaired lung function assessed by the value of forced vital capacity (FVC) and diffusion of lung carbon monoxide (DLCO) at the time of diagnosis, or decline in lung function within 6 or 12 months after the diagnosis, are the best predictive markers of survival but fail to assess or to predict lung function decline. Until recently, lung transplantation was the only IPF treatment and remains associated with high morbidity and mortality. Pirfenidone and nintedanib - anti-fibrotic treatments - are now validated therapies in the management of mild-to-moderate IPF defined by FVC ≥ 50% of predictive value and by DLCO ≥ 30 % of predicted value. Several international clinical trials demonstrated that pirfenidone and nintedanib significantly reduce the lung function decline and the exacerbations incidence and significantly improve survival. The emergence of these innovative but costly therapies - which are associated with a non-negligible rate of adverse effects - requires the development of tools to evaluate their effectiveness and monitor anti-fibrotic activity. The 18-fluorodesoxyglucose (18FDG) lung uptake may be the first tool to predict early therapeutic response. PET offers the possibility to quantify in vivo and non-invasively the cell metabolism, using a non-metabolizable substrate labeled as 18FDG. Several parameters can be measured in an automated and reproducible manner such as the mean uptake intensity (SUV mean), the maximum uptake intensity (SUV max), the metabolic lung volume measurement (MLV) or finally the measurement of tissue glycolytic activity or TLG (total lesion glycolysis). 18FDG PET scanner plays a key role in the diagnosis and monitoring of neoplasia and inflammatory diseases such as sarcoidosis. Recent studies reported a change of the metabolic activity of pulmonary fibroblasts issued from IPF, showing increase of glycolytic activity. In a recent study, the investigators demonstrated a strong correlation between the lung uptake parameters and the lung function tests results and prognostic score GAP. In addition, MLV and TLG were prognostic and independently associated with progression-free survival at 12 months. Preliminary data suggest that the intensity of lung 18FDG uptake may be a prognostic marker but also a predictive marker of response to anti-fibrotic treatments. A prospective study must be conducted to confirm or refute these observations.

Primary objective: The main objective of this study is to describe the changes of 18FDG lung uptake assessed by TLG variation in patients with IPF, 12 weeks after the initiation of pirfenidone.

Secondary objectives: Secondary objectives include the following : 1. To describe the changes of 18FDG lung uptake assessed by other 18FDG indices (SUVmean, SUVmax and MLV) in patients with IPF, 12 weeks after the initiation of pirfenidone ; 2. To study the relationship between the variation of 18FDG lung uptake 12 weeks after the initiation of pirfenidone therapy (as assessed by the changes of TLG, SUVmean, SUVmax and MLV) and the decline of FVC 12, 24, 36 and 48 weeks after the initiation of pirfenidone therapy ; 3. To estimate the predictive performance of the variation of 18FDG lung uptake 12 weeks after the beginning of pirfenidone therapy for therapeutic efficacy at 24 weeks.

Experimental plan: This is an interventional, prospective, multicenter, proof of concept study. 18FDG PET-scanner will be performed at baseline and 12 weeks after the beginning of pirfenidone treatment in each patient. Lung Function Tests will be also performed before and 12 weeks after initiation of pirfenidone treatment and will be repeated every 12 weeks until 48 weeks after pirfenidone initiation. A clinical examination and liver enzymes will be assessed every 12 weeks. The occurrence of any adverse event will be collected throughout the trial. LFTs will be interpreted blindly from the results of 18FDG uptake.

ELIGIBILITY:
Inclusion Criteria:

1. IPF, diagnosed accordingly to ATS/ERS/JRS/ALAT international guidelines
2. FVC≥50% and DLCO≥30%
3. Decision to initiate a treatment with pirfenidone
4. Affiliation to the French social security system

Exclusion Criteria:

Will be non-eligible in this study any patient:

1. with an age lower than 18 years
2. with a life expectancy lower than 12 months as assessed by the investigator
3. taking an anti-fibrotic treatment (pirfenidone, nintedanib or any experimental molecule) in the previous three months
4. treated by corticosteroid therapy (daily dose > 10 mg, prednisone equivalent)
5. with neoplasia localized in thorax
6. with contraindication to pirfenidone according to the French Summary of Product Characteristics : hypersensitivity to the active substance or to any of the excipients, past history of angioedema with pirfenidone, concomitant treatment with fluvoxamine, severe or terminal hepatic insufficiency, severe renal insufficiency (CrCl <30ml / min) or end-stage requiring dialysis
7. with a positive pregnancy test or currently breastfeeding
8. with contraindication to performing a 18FDG PETscan, ie 18FDG hypersensitivity
9. with emphysema extension >15% on HRCT according to Cottin et al (16).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Changes of 18FDG lung uptake (TLG variation) in patients with IPF 12 weeks after the initiation of pirfenidone | 12 weeks
  To describe the changes of 18FDG lung uptake assessed by TLG variation in patients with IPF 12 weeks after the initiation of pirfenidone

SECONDARY OUTCOMES:
Change of 18FDG lung uptake in patients with IPF 12 weeks after the initiation of pirfenidone : variation of SUVmean between baseline and after 12 weeks of treatment | 12 weeks
  Values of SUVmean will be compared between baseline (treatment initiation with pirfenidone) and the 12 weeks using a Wilcoxon's signed rank test
Change of 18FDG lung uptake in patients with IPF 12 weeks after the initiation of pirfenidone : variation of SUVmax between baseline and after 12 weeks of treatment | 12 weeks
  Values of SUVmax will be compared between baseline (treatment initiation with pirfenidone) and the 12 weeks using a Wilcoxon's signed rank test
Change of 18FDG lung uptake in patients with IPF 12 weeks after the initiation of pirfenidone : variation of MLV between baseline and after 12 weeks of treatment | 12 weeks
  Values of MLV will be compared between baseline (treatment initiation with pirfenidone) and the 12 weeks using a Wilcoxon's signed rank test
Variation of the PET parameter SUVmean between baseline and 12 weeks and FVC at 12, 24, 36 and 48 weeks | 48 weeks
  Relationship between the variation of SUVmean values between baseline and 12 weeks after treatment initiation and the decline of FVC over time will be assessed using a linear mixed effect model of the evolution of FVC over time and the effect of the change of each PET parameter on the decline of FVC over time will be tested
Variation of the PET parameter SUVmax between baseline and 12 weeks and FVC at 12, 24, 36 and 48 weeks | 48 weeks
  Relationship between the variation of SUVmax values between baseline and 12 weeks after treatment initiation and the decline of FVC over time will be assessed using a linear mixed effect model of the evolution of FVC over time and the effect of the change of each PET parameter on the decline of FVC over time will be tested
Variation of the PET parameter TLG between baseline and 12 weeks and FVC at 12, 24, 36 and 48 weeks | 48 weeks
  Relationship between the variation of TLG values between baseline and 12 weeks after treatment initiation and the decline of FVC over time will be assessed using a linear mixed effect model of the evolution of FVC over time and the effect of the change of each PET parameter on the decline of FVC over time will be tested
Variation of the PET parameter MLV between baseline and 12 weeks and FVC at 12, 24, 36 and 48 weeks | 48 weeks
  Relationship between the variation of MLV values between baseline and 12 weeks after treatment initiation and the decline of FVC over time will be assessed using a linear mixed effect model of the evolution of FVC over time and the effect of the change of each PET parameter on the decline of FVC over time will be tested
Evaluation of the performance of the PET scanner (Sensitivity, Specificity, Positive predictive value and Negative predictive value) using the variation of each PET parameter and the therapeutic response at 24 weeks (succes versus failure) | 24 weeks
  The performance of the PET scanner (Sensitivity, Specificity, Positive predictive value, and Negative predictive value) will be studied using the variation of each PET parameter and the therapeutic response at 24 weeks.
  A non-parametric Wilcoxon test will be used to compare the variation of each PET parameter according to the therapeutic response.
  The therapeutic response will be classified as therapeutic failure in the case of any of the following events between pirfenidone treatment initiation and 24 weeks: a relative decline in percent predicted FVC ≥10%, an absolute decline in 6MWT distance ≥50 m, or death from any cause, or as therapeutic success (in any other case).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Crestani, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Pneumologie A Centre constitutif de référence des maladies pulmonaires rares Hôpital Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided